CLINICAL TRIAL: NCT03588624
Title: Study of the TearCare System in Dry Eye Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sight Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06001
Record Dates: First submitted 2018-07-03; First posted 2018-07-17 (Actual); Results first posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- TearCare (Experimental): All subjects in the study were successfully treated with the TearCare device and manual expression of their eyelids, one time at the baseline visit.
  Interventions: Device: TearCare

INTERVENTIONS:
Device: TearCare — The TearCare procedure includes the delivery of thermal energy to the external surface of the eyelids for 15 minutes, immediately followed by manual expression of each eyelid.

SUMMARY:
This study was conducted to evaluate the short-term (1 month) safety and effectiveness of a single TearCare procedure to treat adult patients with dry eye disease.

DETAILED DESCRIPTION:
This was a prospective, single-arm, post-market, exploratory treatment study designed to collect clinical data regarding the safety and effectiveness of the TearCare System. To reduce potential bias in the study, study staff performing the endpoint assessments was independent of the clinician performing the TearCare procedure.

In this study, all subjects received the TearCare procedure. The TearCare procedure included an in-office 15 minute treatment session with the TearCare System immediately (i.e. within 3 minutes) followed by manual expression of the meibomian glands using the Express Forceps. Subjects received one in-office TearCare procedure at the baseline visit and then had follow-up visits at 1 week and 1 month.

This study was conducted at 3 sites in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. At least 22 years of age
2. Reports dry eye symptoms within the past 3 months
3. Reports having to use artificial tears or lubricants regularly over the past month to relieve dry eye symptoms.
4. OSDI Score of ≥23
5. TBUT of ≤7 seconds in both eyes
6. Meibomian gland obstruction in both eyes based on a total Meibomian Gland Secretion Score ≤15 in each eye.
7. At least 15 glands in each lower eyelid should be expressible, with a sterile cotton swab, at the slit lamp.
8. Best spectacle corrected visual acuity of 20/100 or better in both eyes.
9. Willing and able to comply with the study procedures and follow-up
10. Willing and able to provide informed consent
11. English-speaking

Exclusion Criteria:

1. Any active, clinically significant ocular or peri-ocular infection or inflammation
2. Recurrent clinically significant eye inflammation, other than dry eye, within 3 months prior to enrollment
3. History of eyelid, conjunctiva or corneal surgery (including refractive surgery) within the past year. In addition, subjects with any history of the following are excluded: chalazion surgery, surgery on the tarsal conjunctiva, radial keratotomy (RK), complicated blepharoplasty, lid reconstruction, or significant complications post-refractive surgery.
4. Any office-based dry eye treatment (e.g. IPL, thermal pulsation [Lipiflow], etc.) within 12 months prior to enrollment. In addition Blephex or debridement within 3 months prior to enrollment is an exclusion.
5. Meibomian gland expression within 6 months prior to enrollment. In addition, any history of meibomian gland probing is an exclusion.
6. In the clinical judgement of the investigator, meibomian glands have significant capping, atrophy, or are unable to be expressed, digitally or with a sterile cotton swab.
7. Contact lens use within the past 2 weeks (Subjects must refrain from wearing contact lenses for the duration of the study.)
8. Use of TrueTear device within the past 2 weeks (Subjects must refrain from using the TrueTear device for the duration of the study.)
9. History of Ocular Herpes Simplex or Ocular Herpes Zoster
10. Clinically significant ocular surface abnormalities that may affect tear film distribution or treatment (e.g. pterygium, anterior membrane dystrophy, etc.)
11. Clinically significant eyelid abnormalities in either eye (e.g. entropion/ectropion, blepharospasm, aponeurotic ptosis, lagophthalmos, notching of lid margin, distichiasis, trichiasis)
12. Clinically significant anterior blepharitis. In addition, collarettes or flakes of more than one quarter of the eyelid are excluded.
13. Clinically significant dermatologic or cutaneous disease of the eyelid or periocular area
14. Ocular trauma within 3 months prior to enrollment
15. Any active, clinically significant allergic, vernal, or giant papillary conjunctivitis
16. Known history of diminished or abnormal facial, periocular, ocular or corneal sensation
17. Corneal surface abnormalities such as corneal epithelial defects (other than punctate staining), ulcers, corneal epithelial dystrophies, keratoconus, and ectatic disease of the cornea
18. Punctal occlusion or punctal plug placement within 30 days prior to enrollment
19. Systemic diseases resulting in dry eye (e.g. autoimmune diseases such as Sjogren's syndrome, rheumatoid arthritis, lupus, Graves' disease, sarcoidosis, etc.)
20. Allergies to silicone tissue adhesives
21. Use of Restasis or Xiidra within 60 days prior to enrollment. Subject must also be willing to remain off these drugs for the duration of the study.
22. Use of antihistamines (oral or topical) within 10 days prior to enrollment. Subject must also be willing remain off antihistamines for the duration of the study.
23. Subject is currently on a systemic medication(s) (other than anti-histamines) that is known to cause ocular dryness (e.g. diuretics, anti-hypertensives, anti-depressants, hormone therapy) and whose dose of this medication(s) has not been stable within 30 days prior to enrollment. There must be no anticipated adjustments to the dose of these medications for the duration of the trial.
24. Subject has taken or is currently taking Accutane
25. Subject requires chronic use (i.e. for any portion of the study) of topical ophthalmic antibiotics, anti-glaucoma medications, steroids, non-steroidal anti-inflammatory medications or who has been on any of these medications within 30 days prior to enrollment
26. Subject is currently using Retin A or Latisse
27. Participation in another ophthalmic clinical trial within one year prior to enrollment. Subject must also be willing to refrain from another ophthalmic study for the duration of the study.
28. Co-existing condition, either ocular or non-ocular that, in the judgement of the investigator could affect the safety or effectiveness of treatment or the compliance of the subject to the protocol. Subjects who are pregnant or nursing or have active, wet macular degeneration are excluded.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2018-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaime C Dickerson, PhD, Study Director — Sight Sciences
Locations (3):
- United States (3):
  - Eye Research Institute, Newport Beach, California
  - Arlington Eye Physicians, Arlington Heights, Illinois
  - Kentucky Eye Institute, Lexington, Kentucky

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- TearCare (Single Procedure): All subjects in the study were successfully treated with the TearCare device and manual expression of their eyelids, one time at the baseline visit.
Period: Overall Study
Arm/Group | TearCare (Single Procedure)
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TearCare (Single Procedure)
Number analyzed (Participants) | 29
Age, Customized [Mean (Inter-Quartile Range); unit: years] | 60.6 [37 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 26
  Hispanic | 3
Region of Enrollment [Number; unit: participants]
  United States | 29
Single TearCare® procedure to treat adult patients with dry eye disease [Count of Participants; unit: Participants] | 29
Tear Break Up Time [Mean (Standard Deviation); unit: seconds] — The TBUT was evaluated by measuring the time to breakup of the tear film following a complete blink when viewed through the slit-lamp using a cobalt blue filter. The TBUT was recorded using a stopwatch for each eye as the average of 3 measurements at each visit. The change in TBUT was The difference between the mean baseline value and the mean Month 1 value. The TBUT for each eye for a subject was averaged. An increase in TBUT represents an improvement.
  seconds | 3.7 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Tear Break-Up Time (TBUT) at 1-month From Baseline
Description: TBUT is an indicator of tear film instability and measures the length of time it takes for the tear film to break down. An increase in TBUT represents an improvement.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | TearCare (Single Procedure)
Number analyzed (Participants) | 29
seconds | 3.1 (2.2)

2. Secondary Outcome: Mean Change in Ocular Surface Disease Index (OSDI) Score From Baseline to Month 1
Description: The Ocular Surface Disease Index (OSDI) questionnaire is a validated questionnaire that consists of 12 questions to assess ocular symptoms, their impact on patient vision-related functioning, and environmental factors triggering the symptoms.
  OSDI Scale Dry Eye Grade 12 or less - Normal 13-22 - Mild 23-32 - Moderate 33 or greater - Severe. Scores may range from 0 (best possible), to 100 (worst possible).
  Mean change from baseline at Month 1 is the difference between the mean score at Month 1 and at baseline. A negative score represents improvement.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | TearCare (Single Procedure)
Number analyzed (Participants) | 29
scores on a scale | 25.8 (24.3)

3. Secondary Outcome: Total Meibomian Gland Secretion Score at 1 Month
Description: The Meibomian Gland Secretion Scoring is an assessment of the quality of the secretions produced by the meibomian glands in the lower eyelids. Fifteen meibomian glands in each of the lower eyelids were gently pressed and the secretions were scored on the scale below. Sum of the grade (0 - 3) for each of the 15 glands. Range for this score is 0-45. A higher number indicates more normal meibomian gland activity.
  Score Description of Secretion 0 Nothing
  1. Toothpaste
  2. Cloudy
  3. Clear
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TearCare (Single Procedure)
Number analyzed (Participants) | 29
score on a scale | 14.4 (7.3)

4. Secondary Outcome: Corneal Staining Score at1 Month
Description: The structural effect of dry eye disease (DED) on subjects' ocular surface and its severity was assessed using corneal and conjunctival staining. The degree of staining was quantified using the NEI/Industry Grading System which scores 5 regions of the cornea and 6 regions of the conjunctiva using a scale from 0 to 3. On this scale, 0 indicates no staining and 3 indicates severe staining. The score for the regions of the cornea were added to obtain a total score that ranged from 0-15 where 0 indicates no ocular surface damage or dry eye.
Time Frame: 1 month
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | TearCare (Single Procedure)
Number analyzed (Participants) | 29
score on a scale | 4.1 (2.8)

5. Secondary Outcome: Conjunctival Staining Score at 1 Month
Description: The structural effect of dry eye disease (DED) on subjects' ocular surface and its severity was assessed using corneal and conjunctival staining. The degree of staining was quantified using the NEI/Industry Grading System which scores 5 regions of the cornea and 6 regions of the conjunctiva using a scale from 0 to 3. On this scale, 0 indicates no staining and 3 indicates severe staining. The score for the regions of the conjunctiva were added to obtain a total score that ranged from 0-18, where 0 indicates no ocular surface damage or dry eye.
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TearCare (Single Procedure)
Number analyzed (Participants) | 29
score on a scale | 4.7 (3.0)

ADVERSE EVENTS:
Time Frame: 1 Month
Arm/Group | TearCare (Single Procedure)
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 2/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TearCare (Single Procedure) (N=29)
Worsening of two or more lines on the Snellen visual acuity (Eye disorders) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-30): https://cdn.clinicaltrials.gov/large-docs/24/NCT03588624/Prot_SAP_000.pdf